CLINICAL TRIAL: NCT02507882
Title: Impact of IL-28B rs12979860 and rs4803217 Gene Polymorphisms Associated With miRNAs Deregulation on HCV-related Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr.Waleed Samir (Other)
Responsible Party: Sponsor-Investigator, Dr.Waleed Samir, Director of Clinical and Research Laboratory& Head of Molecular Biology Unit, Egyptian Liver Hospital, Egyptian Liver Hospital
Organization: Egyptian Liver Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ELH - 2015 - IL28
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: HCV Infection ( Genotype 4)
MeSH Terms: conditions — Hepatitis C

ARMS (3):
- HCC (Experimental): This group will include patients with chronic hepatitis C (no. =135)
  Interventions: Biological: IL28B Polymorphism; Biological: miRNA quantification
- HCC with Cirrhosis (Experimental): This group will include patients with chronic hepatitis C (no. =135) with cirrhosis (F4).
  Interventions: Biological: IL28B Polymorphism; Biological: miRNA quantification
- HCV related HCC patients (Experimental): This group will include patients with HCV related HCC (no. =135) This is confirmed by presence of focal lesion detected by Imaging (computed tomography (CT) and ultrasound), and elevated serum AFP.
  Interventions: Biological: IL28B Polymorphism; Biological: miRNA quantification

INTERVENTIONS:
Biological: IL28B Polymorphism — SNP rs12979860 and 4803217 will be determined in whole blood by allelic discrimination using specific probes by real time PCR.
Biological: miRNA quantification — RNAs will be extracted from serum using miRNeasy Mini Kit (Quiagen) according to the manufacturer's instruction.
  The RNA purity will be assessed by the RNA concentration and quantified by NanoDrop ND-1000 (Nanodrop, United States).
  cDNA will be obtained by miScript II Reverse Transcription Kits (Quiagen) A Preamplification will be performed using miScript PreAMP PCR Kits (Quiagen) Real Time PCRarray will be done using miScript miRNA PCR Arrays, with SYBR Green PCR Master Mix (Quiagen).

SUMMARY:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer deaths worldwide as well as in Egypt. Despite improvements in HCC therapy, the prognosis for HCC patients remains poor. Today molecular, genomic and epigenomic aberrations in tumors are being deeply investigated. Many biomarkers were associated to HCC onset, and they could be useful for clinicians, but all show some limitations and no one is so early to predict the HCC onset.

It is estimated that 51.5% of HCC cases can be attributed to HCV infection. Moreover, there is a large occult reservoir of HCV caused chronic liver disease in approximately 9 % in the Egyptian with estimated 6 million HCV chronic infections and estimated 150 000 new infections per year. Among them, we have to mention the polymorphism of IL28B gene rs12979860 C/T. and rs 4803217. The IL-28B gene encodes interferon-lambda 3 (IFN-λ3), which belongs to the type III IFN family. IFN-λ interacts with a transmembrane receptor inducing a potent antiviral response. In experimental model of HCV type III IFN was able to inhibit viral replication. IL-28B polymorphisms are linked to the efficiency of the inflammatory process during HCV infection, and to the mechanisms that HCV adopts to escape by innate and adaptive immunity.

During the last years, a number of studies have assessed the association between the IL-28B polymorphisms and risk of HCC and liver cirrhosis (LC) occurrence in various populations; however, results obtained are still inconclusive.

Interestingly, some polymorphisms located at the 3' untranslated region (UTR) of IL28B, e.g. rs 4803217, seem to interfere with the binding of miRNA, to date recognized as important post-transcriptional regulators. In the last years miRNAs acquired a growing relevance as potential biomarkers for several diseases including cancer, and many researches are focusing on understanding their role in cancer.

Thus the objectives of the current proposal are to determine through investigating a cohort of 405 patients, whether IL28B rs12979860 and rs4803217 polymorphisms are associated to the risk of HCC in chronic hepatitis C (CHC) patients and, above all, to identify their role as predictor marker of HCC in CHC, when associated to miRNAs modulation. Data obtained by our work could be helpful in HCC diagnosis, thus leading to the improvement of the patients prognosis. The proposed activities are going to be implemented through a partnership us as Egyptian Liver Research Institute and Hospital (ELRIAH)- Dakhlya- Egypt and Non- Egyptian Partners.

DETAILED DESCRIPTION:
Introduction

Hepatocellular carcinoma (HCC) is the third leading cause of cancer deaths worldwide. Despite improvements in HCC therapy, the prognosis for HCC patients remains poor due to a high incidence of recurrence. An improved understanding of the pathogenesis of HCC development would facilitate the development of more effective outcomes for the diagnosis and treatment of HCC at earlier stages.

Currently, molecular alterations in tumors are being scrutinized at a genome-wide scale, covering different dimensions, such as gene expression, epigenetic changes, chromosomal aberrations, and more recently, next generation sequencing. A large number of molecular markers are associated with the development of HCC. that could be useful in the clinic; however, racial differences have been reported, and these need to be examined more thoroughly.

It is estimated that 51.5% of HCC cases can be attributed to HCV infection. Among them, we have to mention the polymorphisms of IL28B gene, e.g. rs12979860 C/T and rs4803217. The IL-28B gene encodes interferon-lamda 3 (IFN-λ3), which belongs to the type III IFN family including IFN-λ1, IFN-λ2, and IFN-λ3. IFN-λ interacting with a trans membrane receptor induces potent antiviral responses mediated by the activation of the JAK-STAT and MAPK pathways. IL-28B polymorphisms are linked to the efficiency of the inflammatory process during HCV infection and to the mechanisms that HCV adopts to escape by innate and adap¬tive immunity. Interestingly, since type III IFN has been found to inhibit both HBV and HCV replication in experimental models, During the last years, a number of studies have assessed the association between the IL-28B polymorphisms and risk of HCC and liver cirrhosis (LC) development in different populations; however, the results are inconsistent and inconclusive. For these reasons, a deep comprehension of the impact of IL28B polymorphisms in HCC occurrence is mandatory.

Interestingly, some polymorphisms located at the 3' untranslated region (UTR) of IL28B, e.g. rs 4803217, seem to interfere with the binding of miRNA, to date recognized as important post-transcriptional regulators.

miRNA, in fact, are small, interfering, non-coding RNA that are 21-30 nucleotides in length, that can promote the modulation of more than 200 mRNAs and are widely associated with human cancers. In the last years miRNA acquired a growing relevance as potential biomarkers for several diseases including cancer.

In particular, the discovery of extracellular miRNA, which are stable in circulation, drives a lot of researchers on their evaluation aiming to the identification of new useful and less invasive diagnostic markers also for HCC.

Objectives

The overall goal is to investigate the Impact of IL-28B rs12979860 and rs4803217 gene polymorphisms associated with miRNAs deregulation on HCV-related hepatocellular carcinoma

Specific Objectives:

1. To determine the association of IL 28B polymorphism(s) with the risk of HCC in chronic hepatitis C patients.
2. To screen a wide panel of miRNAs to uncover the deregulated ones during chronic hepatitis C progression toward HCC
3. To identify an association among IL 28B polymorphism(s) and the major deregulated miRNAs as predictor marker of HCC in chronic hepatitis C patients

Research Approach and Methodology

Patients and methods:

Patients:

This study will include 405 Subjects divided into 3 groups:

Group 1. This group will include patients with chronic hepatitis C (no. =135) Group2. This group will include patients with chronic hepatitis C (no. =135) with cirrhosis (F4).

Group3. This group will include patients with HCV related HCC (no. =135) This is confirmed by presence of focal lesion detected by Imaging (computed tomography (CT) and ultrasound), and elevated serum AFP.

• The basis of the sample size calculation is the following:

* Alpha Feto Protein: ses 41-60% , sp 80-94%
* Prevalence of HCC among HCV infected patients: 5-10%
* Calculation is based on specificity of alpha feto protein at average 87%

A total of 405 cases with average 135 cases /group is required, based on confidence 90 and margin of error 5 %, prevalence of HCC among HCV infected patients 7 %

Methods:

1. Serum α fetoprotein levels were routinely tested in all patients with decompensated cirrhosis. AFP levels were generally elevated in cases that were proved to be HCC, however, the levels ranged from 15 to 650 ng/ml. The diagnosis of HCC was confirmed by a 4 phase multidetector computed tomography (CT) scan or dynamic contrast enhanced magnetic resonance imaging (MRI).
2. HCV RNA quantification. Plasma will be obtained and HCV RNA determined by RT-PCR of plasma using Cobas AmpliPrep/COBAS TaqMan HCV Test (Roche Diagnostics, Branchburg, (NJ).
3. IL28B Polymorphism:

   SNP rs12979860 and 4803217 will be determined in whole blood by allelic discrimination using specific probes by real time PCR.
4. miRNA quantification

   RNAs will be extracted from serum using miRNeasy Mini Kit (Quiagen) according to the manufacturer's instruction.

   The RNA purity will be assessed by the RNA concentration and quantified by NanoDrop ND-1000 (Nanodrop, United States).

   cDNA will be obtained by miScript II Reverse Transcription Kits (Quiagen) A Preamplification will be performed using miScript PreAMP PCR Kits (Quiagen) Real Time PCRarray will be done using miScript miRNA PCR Arrays, with SYBR Green PCR Master Mix (Quiagen).
5. Statistical Analysis:

Statistical analyses will be performed using SPSS Statistics software. P-values, 0.05 were considered significant.

IL28B SNPs comparisons will be done by stratifying patients according to rs12979860CC and rs12979860CT/TT genotypes and 4803217 Analysis miRNA PCR Array will be done by specific Data Analysis Software specifically supplied by Quiagen.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected patients confirmed by RT-PCR with and without fibrosis, cirrhosis and HCC

Exclusion Criteria:

* HCV/HIV co-infection

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
IL-28B rs12979860 and rs4803217 Genotype evaluation | 6 months to 1 year from the start of the study
  Different types of IL28B and their relation to the progressiveness of HCC
Specific miRNA levels and their association with degree of fibrosis, cirrhosis and HCC | 1 to 2 years from the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Liver Hospital, Sherbein, Dakhlya, Egypt

REFERENCES:
- [Result] Doss W, Shiha G, Hassany M, Soliman R, Fouad R, Khairy M, Samir W, Hammad R, Kersey K, Jiang D, Doehle B, Knox SJ, Massetto B, McHutchison JG, Esmat G. Sofosbuvir plus ribavirin for treating Egyptian patients with hepatitis C genotype 4. J Hepatol. 2015 Sep;63(3):581-5. doi: 10.1016/j.jhep.2015.04.023. Epub 2015 May 1. PMID 25937436